CLINICAL TRIAL: NCT01727830
Title: Influence of Hemodilution on Coagulation, pH, Platelet Function, Laboratory Values and ROTEM in Volunteers Using HES 6%, Gelatine and Balanced Gelatine and the Reversal of Coagulopathy With F XIII and Fibrinogen
Brief Title: Hemodilution and Coagulopathy With 3 Colloids
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2012-0042
Record Dates: First submitted 2012-11-05; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Dilutional Coagulopathy
MeSH Terms: interventions — Gelatin; physiogel; In Vitro Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Induced Coagulopathy by HES (Tetraspan), Gelatin (Physiogel), Gelatin balanced (Physiogel balanced) — Blood drawn from volunteers
  Other Names: This trial is in vitro and made with blood of healthy volunteers.; Thus no drug no intervention beside drawing blood is beeing performed.

SUMMARY:
Aim of this in vitro trial is to assess the effect on blood coagulation after 60 % dilution with different colloids (HES 130/0.42, Gelatin and Gelatin balanced) and investigate reversibility by replacement of fibrinogen (FBG), factor XIII (F XIII), and the combination of FBG and FXIII.

In blood of 12 volunteers the following measurements are performed at baseline and 60% dilution with HES 130/0.42, Gelatin or Gelatin balanced: Blood gas analyses, coagulation factor concentrations (F II,F VII,F VIII,F XIII), impedance aggregometry and rotational thrombelastometry (ROTEM®). Then FBG, F XIII and a combination of both was added, in concentrations corresponding to 6 g FBG and 1250 IU F XIII in adults. ROTEM® measurements and determination of factor concentrations are again performed.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* signed informed consent from before blood withdrawal

Exclusion criteria:

* known coagulation disorders,
* any form of anticoagulation therapy,
* use of acetyl-salicylic acid within the past five days,
* use of non-steroidal anti-inflammatory agents within the past 24 hours,
* known renal disease or plasma concentrations of aspartate aminotransferase (>50 U l -1) or alanine aminotransferase (>50 U l-1)
* patients incapable of understanding the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Reversibility of in vitro induced coagulopathy | Same day when blood was drawn
  Coagulopathy in vitro measured after 60 % dilution with HES, Gelatin and Gelatin balanced. Addition of fibrinogen and factor XIII as well as their combination and measurement if the coagulopathy was corrected.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Theusinger, MD, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich, Switzerland